CLINICAL TRIAL: NCT05998044
Title: Effect of Video-based Exercise on Premenstrual Symptoms: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, assistant professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar66
Record Dates: First submitted 2023-08-09; First posted 2023-08-18 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-09

CONDITIONS: Premenstrual Syndrome; Stress
Keywords: stress; Pilates Based Exercises
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: Pilates exercises will be given to the experimental group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Before starting the study for the Control Group, the participants were informed about the research and their consent will be obtained. Afterwards, evaluation surveys will be applied. They will be asked not to participate in any regular exercise for 8 weeks. At the end of 8 weeks, re-evaluation surveys will be applied.
  Interventions: Other: control
- pilates group (Experimental): After people fill out the evaluation questionnaires, they will watch the video recording of pilates based exercises via the link sent to them via Google Drive, and they will be applied twice a week for 8 weeks. All exercises in the video recording will be explained in written, applied and verbal form by the physiotherapist, and they will be asked to practice. Every week, feedback will be received from people that they have done the exercises via their contact numbers. The average application time of the exercises is 30-40 minutes (with the first 10 minutes of warming up and the last 5 minutes of stretching). Participants will be asked to open the video recording each time they exercise and follow them to do the exercises. At the end of 8 weeks, re-evaluation surveys will be applied.
  Interventions: Other: Pilates Based Exercises

INTERVENTIONS:
Other: Pilates Based Exercises — The average application time of the exercises is 30-40 minutes (with the first 10 minutes of warming up and the last 5 minutes of stretching). The first four exercises were used for the warm-up period and the last four exercises were used for the stretching period. The exercises will be done as 1 set of 8 repetitions. The Hundred exercise will be increased to 10 sets of 10 reps every two weeks to 10 reps, 12 reps, and 14 reps, respectively. Participants will be asked to open the video recording each time they exercise and follow them to do the exercises.
  Exercise Program:
  * Arm Circles
  * Toe Touch
  * bridge
  * Shoulder Bridge
  * Chest Lift
  * Hundred
  * Roll Up
  * Leg Circles
  * Chris Cross
  * Side Kick
  * Side Leg Circles
  * one leg kick
  * double leg kick
  * Swan
  * Single leg Stretch
  * Double leg Stretch
  * saw
  * Spine Stretch
  Arms: pilates group
Other: control — They will be asked not to participate in any regular exercise for 8 weeks.
  Arms: control group

SUMMARY:
The aim of this study is to examine the effects of Pilates Based Exercises on premenstrual symptom (PMS) symptoms, perceived stress level and pain intensity.

DETAILED DESCRIPTION:
The research is a quantitative study, and it is in the form of randomized controlled type research, one of the experimental research types. The sample of the study consisted of people who scored above the mild level according to the Premenstrual Syndrome Scale (PMSS) score and volunteered to participate in the study. Participants will be divided into 2 groups as experimental group and control group by randomization method. Sociodemographic Information Form, Premenstrual Syndrome Scale (PMSS), Perceived Stress Scale (PSS) and Mcgill Melzack Pain Scale (MPQ) will be administered to the participants. Pre- and post-intervention data were statistically analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman between the ages of 18-35.
* Not having a condition that prevents exercise (not having orthopedic, cardiopulmonary, mental diseases, etc. that will prevent exercise).
* Not having given birth.
* Volunteer to participate in the study.
* Having a score above the mild level on the PMSS score.
* Normal menstrual cycle.

Exclusion Criteria:

* Having a condition that prevents you from exercising.
* Having a chronic disease.
* Being on any medication regularly.
* Being pregnant.
* Being in the menopausal period.
* Having a gynecological disease (endometriosis, ovarian cyst, pelvic infection, fibroid/uterine tumor etc.)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Premenstrual syndrome is a female-specific disorder.
Enrollment: 50 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
Premenstrual Syndrome Scale (PMSS) | 10 weeks
  PMSS is a 44-item five-point Likert-type scale (Never, Rarely, Sometimes, Often, and Continuous). As stated in the instruction at the beginning of the scale, after the item is read, marking is made by taking into account the scale on the right of the relevant item, according to the "being in the period one week before the period". In scoring the scale, "Never" option is evaluated as 1 point, "Very little" option as 2 points, "Sometimes" option as 3 points, "Often" option as 4 points and "Constantly" option as 5 points. the high score is 220. In addition, PMSS severity classes can be created according to the scores obtained from the scale. Accordingly, a score of 88 and above from the PMSS scale total indicates severe PMS symptoms, and a score below 88 indicates mild premenstrual syndrome symptoms.
Perceived Stress Scale (PSS) | 10 weeks
  The perceived stress scale consists of 14 five-point Likert type items. The scale consists of "never (0), almost never" (1), "sometimes" (2), "often" (3) "very often" (4). In this 14-item form, items 4-5-6-7-9-10 and 13 are scored in reverse. The lowest and highest scores that the participant can obtain from this scale are 0 and 56, respectively. A high total score means a high Perceived Stress Level Scale. It can be said that the participants, whose score range is between 0-35, are in a positive stress level, can effectively cope with stress, and the coping mechanisms they use are also functional. It can be said that the methods used by the participants with a score range of 36-56 to cope with stress are not functional, and therefore they cannot cope with stress effectively.
McGill Melzack Pain Questionnaire (MPQ) | 10 weeks
  MPQ consists of four parts. In the first part, the patient is asked to mark the location of the pain on the body chart and to indicate with the letter 'D' if the pain is deep and 'Y' on the body surface. In the second part, the patient is asked what he compares his pain to. There are 20 word groups with 2 to 6 descriptive words that describe pain in terms of sensory, perceptual and evaluation. The first 10 groups of words include the sensory dimension, the next 5 the perceptual dimension, the 16th group evaluation, and the last 4 groups of multifaceted words that indicate different aspects of pain. In the third part, the relationship of pain with time is asked. In addition, it is asked what reduces pain and what increases it. In the fourth chapter; The patient is asked questions to determine the severity of pain. Evaluation is made on a rating scale consisting of words describing the severity of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyma AYKUT, Study Chair — Uskudar University
Locations (1):
- Üsküdar Unıversıty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dickerson LM, Mazyck PJ, Hunter MH. Premenstrual syndrome. Am Fam Physician. 2003 Apr 15;67(8):1743-52. PMID 12725453
- [Background] Citil ET, Kaya N. Effect of pilates exercises on premenstrual syndrome symptoms: a quasi-experimental study. Complement Ther Med. 2021 Mar;57:102623. doi: 10.1016/j.ctim.2020.102623. Epub 2020 Nov 24. PMID 33246104
- [Background] El-Lithy A, El-Mazny A, Sabbour A, El-Deeb A. Effect of aerobic exercise on premenstrual symptoms, haematological and hormonal parameters in young women. J Obstet Gynaecol. 2015 May;35(4):389-92. doi: 10.3109/01443615.2014.960823. Epub 2014 Oct 3. PMID 25279689
- [Background] Di Lorenzo CE. Pilates: what is it? Should it be used in rehabilitation? Sports Health. 2011 Jul;3(4):352-61. doi: 10.1177/1941738111410285. PMID 23016028
- [Background] Cruz-Ferreira A, Fernandes J, Laranjo L, Bernardo LM, Silva A. A systematic review of the effects of pilates method of exercise in healthy people. Arch Phys Med Rehabil. 2011 Dec;92(12):2071-81. doi: 10.1016/j.apmr.2011.06.018. Epub 2011 Oct 24. PMID 22030232